CLINICAL TRIAL: NCT02587312
Title: Evaluation of Very Low Nicotine Content Cigarettes in Adolescent Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rachel N Cassidy, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1K01CA189300 (NIH)
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Normal Nicotine Content Cigarettes (Active Comparator): SPECTRUM cigarette: 0.8 mg nicotine with 10.5 mg tar (standard nicotine and tar yields of commercially available cigarettes; control condition)
  Interventions: Other: Standard nicotine content cigarettes
- Very Low Nicotine Content Cigarettes (Experimental): SPECTRUM cigarette: 0.03 mg nicotine with 9 mg tar
  Interventions: Other: Very low nicotine content cigarettes

INTERVENTIONS:
Other: Very low nicotine content cigarettes
  Arms: Very Low Nicotine Content Cigarettes
Other: Standard nicotine content cigarettes
  Arms: Normal Nicotine Content Cigarettes

SUMMARY:
The purpose of this study is to determine how reducing the level of nicotine in cigarettes may affect adolescent smoking behavior. In this study, the researchers will randomize adolescent (age 15-19) daily smokers to either receive VLNC cigarettes or normal-nicotine content (NNC) study cigarettes for three weeks following a one-week usual-brand baseline period. Participants will be instructed to smoke only those cigarettes. The researchers will conduct daily assessments of total cigarette use (both study cigarette and non-compliant use of usual brand cigarettes), craving, and withdrawal, weekly assessments of breath carbon monoxide (CO) levels, cigarette acceptability, risk perceptions of VLNC and NNC cigarettes and demand for usual-brand cigarettes, and pre- vs. post-use measures of nicotine and toxicant exposure. Overall, the project will help determine how VLNC cigarettes may affect real-world smoking behavior in adolescents, and illuminate the potential mechanisms through which these products may effect such changes. Such knowledge will contribute to the science base that may inform future policy decisions.

ELIGIBILITY:
Inclusion Criteria:

* current daily smoking (1 or more cigarettes per day for the past 6 months or longer). Participants must meet a breath carbon monoxide criterion of 6 ppm or higher; if this is not met, urine cotinine levels, detected by a NicAlert cotinine screening device, must indicate recent smoking (level 3 or higher).
* Participants must speak and comprehend English well enough to complete study procedures.

Exclusion Criteria:

* Current pregnancy
* Self-reported daily use of alcohol or other non-prescribed drugs (excluding marijuana).
* Participants who are seeking treatment for their smoking or who report that they intend to quit smoking within the next 30 days and have made a 24-hour quit attempt in the past year
* Participants who report current suicidal ideation on the MINI suicide subscale questions 4 & 5 ("In the past month did you have a suicide plan?" and "In the past month did you attempt suicide?"), as well as participants who indicate that they have made a suicide attempt in their lifetime
* Participants who report use of other non-cigarette tobacco products more than 9 out of the last 30 days

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Number of cigarettes smoked per day | End of 3-week intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States